CLINICAL TRIAL: NCT01284660
Title: Docosahexaenoic Acid (DHA) Effects on Cognitive Function, Craving and Psychosocial Factors in Heavy Cigarette Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 00009-11 HYMC
Record Dates: First submitted 2011-01-18; First posted 2011-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: HEAVY TOBACCO SMOKERS

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I. DHA (Active Comparator): Oral ingestion 5 tablets DHA + EPA (daily ingestion DHA 2040 mg and EPA 2710 mg)- (Omega 3 - 950,the Solgar Pharmaceutical Co., Israel).
  Interventions: Dietary Supplement: DHA
- II. Placebo (Placebo Comparator): Oral ingestion of 5 tablets containing the following: gelatin,glycerine,water and soy oil made by the Solgar Pharmaceutical Co., Israel
  Interventions: Dietary Supplement: Oral ingestion of 5 placebo tablets

INTERVENTIONS:
Dietary Supplement: DHA — DHA ingested orally by heavy smokers
  Arms: I. DHA
Dietary Supplement: Oral ingestion of 5 placebo tablets — Oral ingestion of 5 tablets containing the following: gelatin,glycerine,water and soy oil made by the Solgar Pharmaceutical Co., Israel
  Arms: II. Placebo

SUMMARY:
The purpose of this study is to assess effects of Docosahexaenoic Acid (DHA) as an add-on novel supplement on quality of life, cognitive function, craving and psychosocial factors in heavy cigarette smokers. In humans, no previous randomized, double blind controlled study has been conducted to evaluate these effects. The aim of the study is to 1. Test Docosahexaenoic Acid (DHA) beneficial effects on objective clinical indicators of cognitive function (choice reaction time, decision making, impulsivity, facial recognition) in smokers 2. Improvement of quality of life, cigarette craving, psychosocial factors and self-perceptions in smokers treated with DHA supplement

ELIGIBILITY:
Inclusion Criteria:

* Nicotine dependence
* Smoked at least 10 cigarettes per day for the past 12 months and not interested in quitting

Exclusion Criteria:

* Serious kidney, lun, neurological and cardiovascular diseases
* Suicide risk, acute psychosis, severe depression, organic brain syndromes
* Dependence on psychoactive substances other than nicotine

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Reduction in smoking urges and craving | One and a half years
  Reduction in smoking urges and craving to be measured by the following: smoking urges and craving scales; choice reaction time, impulsivity computerized test, quality of life questionnaire, depression inventory, general health questionnaire, scale of perceived social support, facial expression task, self-esteem diary

CONTACTS AND LOCATIONS:
Locations (1):
- Bar Ilan University, Ramat Gan, Israel